CLINICAL TRIAL: NCT01875913
Title: The Power of Curiosity
Brief Title: The Power of Curiosity: Leveraging Curiosity to Motivate People to Complete Health Risk Assessments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Responsible Party: Principal Investigator, Todd Rogers, Professor Todd Rogers, Harvard University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: F24176-101
Record Dates: First submitted 2013-06-07; First posted 2013-06-12 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Intention; Exploratory Behavior
Keywords: Curiosity; Intention; Follow Through
MeSH Terms: conditions — Exploratory Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Message (Experimental): Participants will receive email messages that encourage them to complete their VHR.
  Interventions: Behavioral: Standard Message
- Curiosity Message (Experimental): Participants receive email messages containing "curiosity-inducing" questions. The messages tell the participants that they will receive the answer to the question after they complete their VHR.
  Interventions: Behavioral: Curiosity Message

INTERVENTIONS:
Behavioral: Curiosity Message — Participants will receive email messages that contain one of 8 curiosity-inducing questions. The message will tell participants that they will receive a message with the answer after they complete their VHR (health review that can be completed online).
  Arms: Curiosity Message
Behavioral: Standard Message — Participants will receive email messages that contain "standard" language encouraging them to complete their VHRs (health review that can be completed online).
  Arms: Standard Message

SUMMARY:
The investigators will work with one of Vitality's partner corporations to test whether curiosity can motivate employees to follow through on their virtuous intentions and complete their annual health risk assessment (VHR). Employees will receive email messages that contain either a curiosity-inducing question or a standard encouragement message. The investigators predict that presenting people with curiosity-arousing questions will make them more likely to complete a health risk assessment, as compared to standard messages.

DETAILED DESCRIPTION:
The vast majority of adults express the desire and intention of engaging in healthy behaviors-exercising, losing weight, getting a colonoscopy-but then fail to do so. This has massive individual and societal costs. This research tests a promising intervention to increase the likelihood that an adult will follow through on their health-related intentions. Curiosity can be a powerful motivator and can cause people to engage in new behaviors (Tomkins 1962; Silvia 2006); however, curiosity has not yet been used as an intervention to help people follow-through on their intentions. In this project, the investigators target employees who have failed to complete their annual Vitality Health Review (VHR) and test whether curiosity can be used to induce the employees to complete their VHR. The VHR is a medical questionnaire that can help individuals understand medical risk factors they may be prone to. The investigators provide employees with a question and inform them that they will see the answer upon completion of their VHR. The investigators hypothesize that the curiosity-inducing messages will cause employees to follow through on their intention to complete their VHR.

ELIGIBILITY:
Inclusion Criteria:

* Employees at Vitality's partner's worksites that are in Vitality database
* Must have email address on file

Exclusion Criteria:

* Employees that have already completed their VHR by June 11, 2013

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10095 (Actual)
Dates: Start 2013-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Completion of VHR | Measured one month after first message (July 12, 2013)
  Whether the participant completes his/her VHR or not

OTHER OUTCOMES:
Previous VHR Completion during 2012-2013 | On or before July 12, 2013
  Whether employee completed their VHR the previous year
Social Atmosphere at Worksite | On or before August 12, 2013
  Measured by post-intervention survey with questions about how frequently employees at worksite interact and discuss non-work and Vitality-related matters
Curiosity Type | On or before July 12, 2013
  For participants who receive "curiosity" messages, indicates which curiosity message they received.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Rogers, PhD, Principal Investigator — Harvard University; Erin Frey, Principal Investigator — Harvard University
Locations (1):
- Harvard Kennedy School, Cambridge, Massachusetts, United States